CLINICAL TRIAL: NCT03541512
Title: Remote Mindfulness-Education Intervention for Women with Provoked Localized Vulvodynia: a Randomized Clinical Study
Brief Title: Remote Mindfulness Education PLV
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Catherine M Leclair, MD, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18191
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Provoked Localized Vulvodynia
Keywords: Mindfulness therapy; Vulvodynia; Vulvar pain
MeSH Terms: conditions — Vulvodynia | interventions — Mindfulness; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness & Education (Active Comparator): Mindfulness practice using guided HeadSpace medications plus educational materials
  Interventions: Behavioral: Mindfulness + Education
- Education only (Active Comparator): Educational materials only
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Mindfulness + Education — Women in the mindfulness + education group will be asked to meditate daily, 10 minutes a day for the first 4 weeks with the option to increase their time to 20 minutes daily during the second 4 weeks. Women will also receive educational materials each week addressing different themes such as; "Introduction and Overview", "The Vulva", "Provoked Localized Vulvodynia (PLV)", "Treatment of PVL", "The Pelvic Floor", "Sexuality", "Chronic Pain", and "Promoting Sexual Health".
  Other Names: Mindfulness group
  Arms: Mindfulness & Education
Behavioral: Education — Women will also receive educational materials each week addressing different themes such as; "Introduction and Overview", "The Vulva", "Provoked Localized Vulvodynia (PLV)", "Treatment of PVL", "The Pelvic Floor", "Sexuality", "Chronic Pain", and "Promoting Sexual Health".
  Other Names: Education group
  Arms: Education only

SUMMARY:
This is a study designed to learn more about the use of an online remote education and mindfulness practice program for the pain and anxiety associated with provoked localized vulvodynia.

DETAILED DESCRIPTION:
The purpose of study is to evaluate the effectiveness of a remotely delivered mindfulness intervention combined with education for the treatment of the pain and distress associated with Provoked Localized Vulvodynia (PLV). Women with PLV will be randomized to either an app- based mindfulness program (Headspace®) with online education or online education only. Pain and sexual distress with be evaluated through a number of measures. The primary outcome of the study will be the change in distress relating to sexual activity over the 8-week intervention period, which will be measured by a change (reduction) in the Female Sexual Distress Scale (FSDS). Participants will additionally perform a weekly Tampon Test and fill out a weekly survey regarding their perceived pain as well as the frequency of use and completion of the weekly education materials

ELIGIBILITY:
Inclusion Criteria:

* Reported dyspareunia for at least 3 months in non-pregnant, healthy women over aged 18 years old and estrogen replete with confirmed diagnosis of provoked localized vulvodynia (PVL) or positive Q-tip test, meeting Friedrich's criteria for PLV.
* Ability to insert a regular Tampax® tampon
* Phone access
* Cellular phone with ability to download applications
* Reliable Internet Access

Exclusion Criteria:

* Pregnancy
* Active sexual counseling or mindfulness training (within 6 months of study)
* Any other clinical reason for dyspareunia (endometriosis pain, chronic pelvic pain, vulvar dermatoses such as psoriasis, lichen sclerosus, etc).
* Unable or unwilling to complete baseline assessments or agree to be randomized.
* Non-English speaking, as Headspace® is not validated in other languages
* Actively engaged in a meditative practice

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Female Sexual Distress Scale (FSDS) at 8 weeks | Baseline & 8 weeks
  The change in distress relating to sexual activity, measured by a change in the FSDS from baseline (study enrollment) survey. Participants will complete a Female Sexual Distress Scale (FSDS) survey to rate their feelings associated with sexual activities. Survey questions are on a number scale of 0 (Never) to 4 (Always). The FSDS surveys will be completed at baseline and 8 weeks after study enrollment.

SECONDARY OUTCOMES:
Change in Tampon Test Pain Scores at 8 weeks | Baseline & 8 weeks
  The change in tampon test pain scores (a validated tool that measures introital pain). The tampon test is a validated tool used to measure (vulva) vestibular skin pain by having participants insert and remove a tampon. Participants will be asked to rate their pain along a 100 mm Visual Analog Scale on a scale of 0 (No pain) to 10 (pain as bad as you can imagine). This test will occur at baseline and 8 weeks after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Leclair, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No